CLINICAL TRIAL: NCT05981950
Title: Real-world Application of Using Artificial Intelligence in Diagnosing Retinal Diseases
Brief Title: Real-world of AI in Diagnosing Retinal Diseases
Status: Recruiting | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Wenbin Wei, Prof, Beijing Tongren Hospital
Other Study IDs: Real-world RAIDS
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Artificial Intelligence; Retinal Diseases
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retinal diseases diagnosed by artificial intelligence algorithm: An artificial intelligence algorithm was applied to diagnose referral diabetes retinopathy, referral age-related macular degeneration, referral possible glaucoma, pathological myopia, retinal vein occlusion, macular hole, macular epiretinal membrane, hypertensive retinopathy, myelinated fibers, retinitis pigmentosa and other retinal lesions from fundus photography.
  Interventions: Diagnostic Test: artificial intelligence algorithm

INTERVENTIONS:
Diagnostic Test: artificial intelligence algorithm — Retinal diseases diagnosed by artificial intelligence algorithm

SUMMARY:
The objective of this study is to apply an artificial intelligence algorithm to diagnose multi-retinal diseases in real-world settings. The effectiveness and accuracy of this algorithm are evaluated by sensitivity, specificity, positive predictive value, negative predictive value, and area under curve.

DETAILED DESCRIPTION:
The objective of this study is to apply an artificial intelligence algorithm to diagnose referral diabetes retinopathy, referral age-related macular degeneration, referral possible glaucoma, pathological myopia, retinal vein occlusion, macular hole, macular epiretinal membrane, hypertensive retinopathy, myelinated fibers, retinitis pigmentosa and other retinal lesions from fundus photography. tic 45-degree fundus cameras, trained operators took binocular fundus photography on participants. Operators were then asked to identify gradable images and unload for algorithm diagnosis. The effectiveness and accuracy of this algorithm are evaluated by sensitivity, specificity, positive predictive value, negative predictive value, area under curve, and F1 score.

ELIGIBILITY:
Inclusion Criteria:

* fundus photography around 45° field which covers optic disc and macula
* complete identification information

Exclusion Criteria:

* insufficient information for diagnosis

Ages: 1 Year to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population is derived from an anonymous database that contains health examination results of the general population.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
Area under curve | 1 month
  We used the receiver operating characteristic (ROC) curve and area under curve to examine the ability of this artificial intelligence algorism recognition and classification of retinal diseases.
Sensitivity and specificity | 1 month
  We used sensitivity and specificity to examine the ability of this artificial intelligence algorism recognition and classification of retinal diseases.
Positive predictive value, negative predictive value | 1 month
  We used positive predictive value and negative predictive value to examine the ability of this artificial intelligence algorism recognition and classification of retinal diseases.
F1 score | 1 month
  We used F1 score to examine the ability of this artificial intelligence algorism recognition and classification of retinal diseases.

CONTACTS AND LOCATIONS:
Locations (1):
- Wen-Bin Wei, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No